CLINICAL TRIAL: NCT06579703
Title: Ketorolac Dosing for Acute Vaso-Occlusive Crisis in Pediatric Patients With Sickle Cell Disease
Brief Title: Ketorolac for Acute Vaso-Occlusive Crisis in Pediatric Sickle Cell Disease
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Blood and Cancer Center at Dell Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Chang_pain in SCD
Record Dates: First submitted 2024-07-24; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Sickle Cell Disease; Sickle Cell Crisis; Veno-occlusive Disease
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Intervention Model Description: Randomized to 1 of 2 arms, parallel dosing
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator, subject, bedside nurse and provider assessing at the bedside will be blinded. There will be an unblinded personnel for dose preparation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Reduced dose Ketorolac Arm A (Experimental): a reduced dose of Ketorolac, 15 mg/mL
  Interventions: Drug: Ketorolac
- Standard of care dose Ketorolac Arm B (Active Comparator): standard of care dose of Ketorolac, 30mg/mL
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — Randomized to a single dose of:
  Arm A: 15 mg/mL (per mL) Arm B: 30 mg/mL (per mL)
  Other Names: Toradol

SUMMARY:
Pediatric patients who present with acute vaso-occlusive pain crisis may have equivalent pain reduction scores at lower dosing of intravenous Ketorolac compared to standard dosing of 0.5 mg/kg/dose IV (<16yo max 15mg, >16yo max 30mg) x 1 dose.

DETAILED DESCRIPTION:
Sickle Cell Disease is characterized by a point mutation that causes red cell polymerization and clinically results in pain events, called vaso-occlusive crises (VOC), and end organ damage. VOC is the most common reason for hospital admissions and ER visits in the SCD population. Ketorolac is an NSAID class medication widely used for pain. Ketorolac reversibly inhibits cyclooxygenase-1 and cyclooxygenase-2 and inhibits the formation of prostaglandins and thromboxane. Specifically, in the SCD pediatric population, Ketorolac was shown to provide adequate pain relief without the need for additional IV analgesics in 50% of patients presenting to the emergency department with VOC. Despite its potential benefits, adverse effects from Ketorolac at standard dosing include gastrointestinal hemorrhage, nephrotoxicity and drug-drug interactions, some of which are dose-dependent. Patients with SCD may be particularly vulnerable to acute kidney injury from nephrotoxic medications given the propensity for chronic kidney disease from ongoing anemia, hemolysis and inflammation. A retrospective review in hospitalized patients with SCD who received at least one dose of ketorolac found that higher doses of ketorolac was a risk factor for acute kidney injury. In addition, a case report on a pediatric patient with SCD showed irreversible renal failure and bleeding complications after administration of ketorolac, despite adequate hydration. The American Society of Hematology guidelines for management of acute and chronic pain in patients with sickle cell disease recommend a short course of NSAIDs in addition to opioids for acute pain management based on very low certainty of evidence.

Several adult studies have suggested that the efficacy of ketorolac analgesia at 10mg is equivalent to higher doses (15mg-90mg) for treatment of various pain syndromes in the ED setting, post-operative and cancer pain. However, these studies excluded patients with SCD whose pain mechanism and pain thresholds may differ from these populations.

The investigators propose a prospective, randomized, double blind clinical trial that will take place in the DCMC Emergency Department and Children's Blood and Cancer Center Hematology Outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with sickle cell disease (any genotype) who present to DCMC Emergency department or outpatient hematology clinic with acute pain.

Exclusion Criteria:

* Patients receiving NSAID medication <6 hours from presentation
* known kidney injury
* sickle nephropathy
* bleeding concerns
* allergy to NSAID medication
* chronic pain patient
* hemodynamic instability as defined by the treating provider

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
FACES Pain Scale-Revised(FPS-R) | Assessed before dose of pain medication and 30 minutes post-dose
  Has a range from 0 to 10 possible. 0 to 3 mild pain, 4 to 6 moderate pain, 7 to 10 severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Chang, MD, Principal Investigator — Director, Comprehensive Sickle Cell Center

REFERENCES:
- [Background] Brandow AM, Carroll CP, Creary S, Edwards-Elliott R, Glassberg J, Hurley RW, Kutlar A, Seisa M, Stinson J, Strouse JJ, Yusuf F, Zempsky W, Lang E. American Society of Hematology 2020 guidelines for sickle cell disease: management of acute and chronic pain. Blood Adv. 2020 Jun 23;4(12):2656-2701. doi: 10.1182/bloodadvances.2020001851. PMID 32559294
- [Result] Shapiro BS. The management of pain in sickle cell disease. Pediatr Clin North Am. 1989 Aug;36(4):1029-45. doi: 10.1016/s0031-3955(16)36735-9. PMID 2666928
- [Result] Jones SF, O'Donnell AM. Clinical pharmacology: traditional NSAIDs and Jones SF, O'Donnell AM. Clinical pharmacology: traditional NSAIDs and selective COX-2 inhibitors. In: Macintyre PE, Walker SM, Rowbotham DJ, et al, eds. Clinical Pain Management (Acute Pain). 2nd ed. London, England: Hodder & Stoughton Limited; 2008:79.
- [Result] Motov S, Yasavolian M, Likourezos A, Pushkar I, Hossain R, Drapkin J, Cohen V, Filk N, Smith A, Huang F, Rockoff B, Homel P, Fromm C. Comparison of Intravenous Ketorolac at Three Single-Dose Regimens for Treating Acute Pain in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2017 Aug;70(2):177-184. doi: 10.1016/j.annemergmed.2016.10.014. Epub 2016 Dec 16. PMID 27993418
- [Result] Staquet MJ. A double-blind study with placebo control of intramuscular ketorolac tromethamine in the treatment of cancer pain. J Clin Pharmacol. 1989 Nov;29(11):1031-6. doi: 10.1002/j.1552-4604.1989.tb03274.x. PMID 2689472
- [Result] Minotti V, Betti M, Ciccarese G, Fumi G, Tonato M, Del Favero A. A double-blind study comparing two single-dose regimens of ketorolac with diclofenac in pain due to cancer. Pharmacotherapy. 1998 May-Jun;18(3):504-8. PMID 9620101
- [Result] Brown CR, Moodie JE, Wild VM, Bynum LJ. Comparison of intravenous ketorolac tromethamine and morphine sulfate in the treatment of postoperative pain. Pharmacotherapy. 1990;10(6 ( Pt 2)):116S-121S. PMID 2082307
- [Result] Simckes AM, Chen SS, Osorio AV, Garola RE, Woods GM. Ketorolac-induced irreversible renal failure in sickle cell disease: a case report. Pediatr Nephrol. 1999 Jan;13(1):63-7. doi: 10.1007/s004670050565. PMID 10100293
- [Result] Baddam S, Aban I, Hilliard L, Howard T, Askenazi D, Lebensburger JD. Acute kidney injury during a pediatric sickle cell vaso-occlusive pain crisis. Pediatr Nephrol. 2017 Aug;32(8):1451-1456. doi: 10.1007/s00467-017-3623-6. Epub 2017 Feb 25. PMID 28238158